CLINICAL TRIAL: NCT06267768
Title: The Effects of Different Inspiratory Pressures on the Diaphragmatic Thickness Fraction and Sternocleidomastoid Muscle Activation in People After Stroke
Brief Title: The Effects of Inspiratory Pressures on Diaphragmatic Contraction in People After Stroke
Status: Completed | Type: Observational
Sponsor: Hong Kong Metropolitan University (Other)
Collaborators: Shenzhen Second People's Hospital (Other)
Responsible Party: Principal Investigator, LIU FANG, PhD student, Hong Kong Metropolitan University
Other Study IDs: REC Reference No.:HE-OT2023/13; Proj.Ref.No.: 2023/3007-R7052 (Other Grant/Funding Number: Research Donation Fund, Hong Kong Metropolitan University)
Record Dates: First submitted 2024-02-04; First posted 2024-02-20 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Stroke
Keywords: Stroke; Diaphragmatic thickening fraction; Sternocleidomastoid muscles; Inspiratory pressures
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke participants: People diagnosed with stroke and meeting all inclusion criteria will be included in this study.
  Interventions: Diagnostic Test: Various intensities of inspiratory muscle training
- Healthy participants: Healthy adults meeting all inclusion criteria will be included in this study.
  Interventions: Diagnostic Test: Various intensities of inspiratory muscle training

INTERVENTIONS:
Diagnostic Test: Various intensities of inspiratory muscle training — Each participant will be asked to perform the lung function test to measure the maximal inspiratory pressure (MIP) after including the study. After the baseline measurement, all participants will be requested to use a nose clip to hold the nose and breathe with the mouth through a pressure threshold inspiratory loading device (POWERbreathe, KH2, England). The inspiratory pressure will be set at 30%, 40%, 50%, 60%, 70%, or 80% of their MIP, in random order. Each MIP intensity protocol consists of 10 breaths. Resting will be allowed between different protocols of contraction intensity (% MIP). During the test, sternocleidomastoid muscle activity will be measured with surface electromyography (sEMG) and diaphragm thickness will be used to assessed with ultrasonography.

SUMMARY:
This is a cross-sectional study to determine the optimal inspiratory muscle training (IMT) intensity for stroke survivors. Participants will breathe through a pressure threshold inspiratory loading device with varying loads in random order. Each IMT intensity protocol consists of 10 breaths. During the test, accessory inspiratory muscle activity will be measured with surface electromyography (sEMG) and diaphragm thickness will be used to assessed with ultrasonography. Repeated-measures ANOVA will be used for statistical analysis to determine the most effective training intensity for future study.

ELIGIBILITY:
Recruitment of participants after a stroke:

The inclusion criteria are:

* clinical diagnosis of ischemic and/or hemorrhagic stroke.
* age ≥ 18 years.
* duration of stroke ranges from 1 month to 12 months after diagnosis.
* had no facial palsy, which could prevent proper labial occlusion.
* had not undergone thoracic or abdominal surgery.
* could understand and follow the verbal instruction.
* stable cardiac conditions.
* no previous history of respiratory problems.

The exclusion criteria are:

* acute myocardial infarction or acute heart failure.
* acute pain on chest or abdominal.
* with the clinical signs of significant pulmonary disease.
* consciousness impaired.
* patient with nasal feeding tube, tracheal tube and/or any condition, which prevent the measurement or training.

Recruitment of healthy participants:

The inclusion criteria are:

* age ≥ 18 years.
* had not undergone thoracic or abdominal surgery.
* no previous history of respiratory problems.

The exclusion criteria are:

* acute myocardial infarction or acute heart failure.
* acute pain in the chest or abdominal.
* with the clinical signs of significant pulmonary disease.
* unstable hypertension, arrhythmias, or unstable cardiovascular conditions, such as fluctuations in blood pressure and heart rate, indicate poor cardiac prognosis or the need for vasopressor medications.
* pregnant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People after stroke and healthy adults
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2024-03-02 (Actual); Primary Completion 2024-08-17 (Actual); Study Completion 2024-08-17 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic thickening fraction | Data will be measured at baseline and at the end of each inspiratory muscle training intensity protocol;
  Diaphragmatic thickening fraction is determined by "(thickness of the diaphragm at end inspiratory - thickness at end expiratory)/thickness at end expiratory". Diaphragmatic thickness will be measured by ultrasonography.

SECONDARY OUTCOMES:
Muscle activation of the sternocleidomastoid muscle | Data will be measured at baseline and at the end of each inspiratory muscle training intensity protocol;
  Surface electromyography will be used to measure accessory inspiratory muscle (sternocleidomastoid muscles) activity during each inspiratory muscle training intensity protocol.
Perceived Exertion Borg scale | Data will be measured at the end of each inspiratory muscle training intensity protocol;
  This is a vertical scale quantified from 0 to 10, where 0 represents no symptoms, and 10 represents the maximum symptoms. The Borg score provides an individual measurement of the exercise intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Tsang William, Principal Investigator — Hong Kong Metropolitan University
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, None Selected, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-29): https://cdn.clinicaltrials.gov/large-docs/68/NCT06267768/Prot_SAP_000.pdf
  • Informed Consent Form (2023-12-29): https://cdn.clinicaltrials.gov/large-docs/68/NCT06267768/ICF_001.pdf